CLINICAL TRIAL: NCT06638177
Title: Obesity and Obesity-Related Factors and Risk of Herpes Zoster and Postherpetic Neuralgia
Brief Title: Obesity and Obesity-Related Factors and Risk of Herpes Zoster (Shingles) and Postherpetic Neuralgia
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sharon G Curhan, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2024P001006
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Herpes Zoster (HZ)
Keywords: shingles; herpes zoster; post-herpetic neuralgia; obesity; plasma metabolomics; observational study
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We have already collected blood from participants. The samples have been stored in liquid nitrogen (-130 degrees C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Health Professionals Follow-Up Study: The HPFS is an ongoing prospective study of 51,529 male health professionals (dentists, veterinarians, pharmacists, optometrists, osteopaths, and podiatrists) who were 40 to 75 years of age at enrollment in 1986. Approximately 97% of participants were of white European descent. Similar to the NHS cohorts, participants have been followed through mailed biennial questionnaires (https://www.hsph.harvard.edu/hpfs/hpfs-questionnaires/) that ascertained medical history, lifestyle, and health-related behaviors, as previously described.88,89 The 2004, 2006, and 2008 questionnaires included questions that elicited information on history of HZ and the year when the episode of HZ occurred. The upcoming 2024 questionnaire will also elicit information on history of HZ, whether participants had been vaccinated against HZ and the date of vaccination.
- Nurses Health Study: In 1976, the NHS I enrolled 121,700 female nurses ages 30 to 55 years who returned a mailed questionnaire regarding their medical history and lifestyle.85,86 There were no exclusions by race; 95% were white reflecting the racial make-up of nurses at that time. Participants receive follow-up questionnaires biennially to record newly diagnosed illnesses and to update lifestyle factors and every 4 years received semiquantitative food frequency questionnaires (FFQs).87 The questionnaires (available at https://nurseshealthstudy.org/participants/questionnaires) are administered every other year, and the 40-year follow-up exceeds 90% of eligible person-time. Information on history of HZ and the date at which HZ occurred was collected on the 2000, 2004, 2008, 2012, 2019, 2021 and 2023 biennial questionnaires. The 2021 and 2023 questionnaires also collected information on whether participants had been vaccinated against HZ and the date of vaccination.
- Nurses Health Study II: In 1989, 116,430 female registered nurses from 15 states ages 25-42 years completed the initial questionnaire and comprise the NHS II. There were no exclusions by race; 2% were black, 2% Asian, and 2% Hispanic. As in NHS I, participants receive follow-up questionnaires biennially (https://nurseshealthstudy.org/participants/questionnaires) to record newly diagnosed illnesses and to update lifestyle factors and every 4 years received semiquantitative food frequency questionnaires.87 The average follow-up rate over 30 years is > 90% of eligible person-time. The 2001, 2005, 2013, 2017, 2019, 2021 and 2023 NHS II questionnaires included questions that elicited information on history of HZ and the year when the episode of HZ occurred. The 2017, 2021 and 2023 questionnaires also collected information on whether participants had been vaccinated against HZ and the date of vaccination.

SUMMARY:
The investigators' objectives are to examine the longitudinal association of obesity and obesity-related factors and risk of incident herpes zoster (HZ), also known as shingles, and the longitudinal association of obesity and obesity-related factors and risk of developing post-herpetic neuralgia (PHN) among those with HZ. The investigators propose to examine more refined assessments of adiposity, leveraging the resources of several large-scale ongoing cohort studies of women and men with decades of follow-up and rich health-related data, including multiple validated anthropomorphic measures, medical history, dietary intake, and lifestyle factors. The investigators will also examine existing data on plasma adipokines, cytokines, and plasma metabolomics. The investigators will use the Nurses' Health Study (NHS I), Nurses' Health Study II (NHS II), and the Health Professionals Follow-up Study (HPFS) (total N>200,000) to prospectively investigate whether obesity and obesity-related factors influence the risk of developing HZ. The investigators have already identified >30,000 cases of incident HZ among the 3 cohorts (reported with high validity) and information on HZ continues to be collected. In addition, the investigators obtained detailed information on HZ course, complications (including PHN), treatment and other related factors on a Zoster Supplemental Questionnaire (ZSQ) administered to those participants in the NHS I and II who reported "shingles" on the main questionnaires (n=10,123 to date). The investigators will also administer the ZSQ to newly identified HZ cases identified on the 2023 NHS I and NHS II biennial questionnaires. No previous study has investigated the longitudinal relation between adiposity and risk of post-herpetic neuralgia (PHN). This study could provide important new insight into how obesity and obesity-related factors influence the risk of HZ, and the risk of developing PHN among individuals with HZ, and how alterations in circulating metabolites and metabolic pathways, including those that are obesity-related, are associated with risk of developing HZ and PHN.

DETAILED DESCRIPTION:
Research Questions: Hypotheses

1. The investigators hypothesize that greater body adiposity is associated with increased risk of developing herpes zoster (HZ). Specifically, the investigators hypothesize that higher body mass index (BMI), larger waist circumference, and higher waist to hip ratio, waist to height ratio, predicted fat mass, predicted percent fat and ABSI are associated with increased risk of developing HZ. The investigators will also examine whether these associations differ by age, sex and other factors.
2. The investigators hypothesize that plasma biomarkers of obesity and of inflammation are independently and longitudinally associated with risk of HZ. Specifically, The investigators hypothesize that lower plasma total and high-molecular-weight (HMW) adiponectin, and higher plasma leptin, IL-6 and CRP are independently associated with higher risk of HZ.
3. The investigators hypothesize that greater body adiposity is associated with increased risk of developing postherpetic neuralgia (PHN). Specifically, The investigators hypothesize that higher body mass index, larger waist circumference, and higher waist to hip ratio, waist to height ratio, predicted fat mass, predicted percent fat and ABSI are associated with increased risk of developing post-herpetic neuralgia (PHN) among those who develop HZ.
4. The investigators hypothesize that obesity-related metabolic dysregulation contributes to HZ risk. Specifically, The investigators hypothesize that circulating levels of metabolites and metabolic pathways that are altered by adiposity and may influence cell-mediated immune function, such as glutamine, arginine, the branched chain amino acids isoleucine, leucine and valine, the tryptophan metabolite kynurenine, and certain fatty acids, such as lysophosphatidylcholines, are associated with risk of developing HZ.
5. The investigators hypothesize that obesity-related metabolic dysregulation contributes to risk of developing PHN among women with HZ. Specifically, the investigators hypothesize that alterations of plasma levels of certain metabolites and metabolic pathways previously implicated in chronic neuroimmune inflammation and increased neurosensitivity, including abnormal fatty acid and amino acid metabolism (e.g. arachidonic acid derived eicosanoids, glutamate-aspartate, tryptophan-kynurenine, and arginine-ornithine metabolic pathways), are associated with the development of PHN among women with HZ.

III. Objectives

A. Objective 1a: To examine whether anthropomorphic measures of obesity from early through middle and later adult life are independently and longitudinally associated with risk of HZ. The investigators will use information on BMI, waist circumference, hip circumference, predicted fat mass and percent fat, ABSI and HZ that has been longitudinally collected across the lifespan among >200,000 women and men. WThe investigators e hypothesize that higher body mass index (BMI), larger waist circumference, higher waist to hip ratio, higher waist to height ratio, higher predicted fat mass, predicted percent fat and ABSI are associated with increased risk of developing HZ. The investigators will also examine whether these associations differ by age, sex and other factors.

B. Objective 1b: To examine whether plasma biomarkers of obesity, the immunomodulatory adipokines leptin and adiponectin, and markers of inflammation, interleukin-6 (IL-6) and C-reactive protein (CRP), are independently and longitudinally associated with risk of HZ. Using existing plasma biomarker information from >19,000 participants, including over 2,500 that developed HZ after the time of the blood collection (incident HZ), the investigators will examine associations of these plasma biomarkers and risk of developing HZ, and examine whether the proposed association between obesity and HZ risk is mediated through immunomodulatory adipokines or inflammation. The investigators hypothesize that lower total and high-molecular-weight (HMW) adiponectin, and higher plasma leptin, IL-6 and CRP are independently associated with higher risk of HZ.

C. Objective 1c: To investigate whether anthropomorphic measures of obesity are associated with higher risk of developing postherpetic neuralgia (PHN) among women with HZ. In a substudy of over 10,000 NHS I and NHS II participants who reported a history of "shingles," the investigators collected detailed information on HZ course, treatment and related complications on a Zoster Supplemental Questionnaire (ZSQ). Information on PHN was validated by medical record review. The investigators hypothesize that higher body mass index, larger waist circumference, and higher waist to hip ratio, waist to height ratio, predicted fat mass, predicted percent fat and ABSI are associated with increased risk of developing PHN.

D. Objective 2a: To assess how obesity-related metabolic dysregulation contributes to HZ risk.

The investigators will conduct an agnostic analysis to identify individual metabolites and metabolic pathways associated with obesity among >13,000 women and men for whom the investigators have comprehensive information on plasma metabolomics profiles. The investigators hypothesize that circulating levels of metabolites and metabolic pathways that are altered by body adiposity and may influence cell-mediated immune function, such as glutamine, arginine, the branched chain amino acids isoleucine, leucine and valine, the tryptophan metabolite kynurenine, and certain fatty acids, such as lysophosphatidylcholines, are associated with risk of developing HZ. The investigators will create a metabolite-based obesity score and assess the degree to which the association between obesity and HZ risk is mediated by the metabolite-based obesity score. Secondarily, the investigators will conduct an agnostic investigation to identify individual metabolites and metabolic pathways associated with risk of developing HZ.

E. Objective 2b: To assess how obesity-related metabolic dysregulation contributes to risk of developing postherpetic neuralgia (PHN) among women with HZ. Among participants who had HZ and completed the Zoster Supplementary Questionnaire (ZSQ) that collected additional details about HZ course, complications and treatment, and for whom information on metabolomics information is available (n=1,005 to date), the investigators will assess the degree to which the potential association between obesity and PHN risk is mediated by the metabolite-based obesity score (developed in Aim 2a above). Secondarily, the investigators will conduct an agnostic investigation to identify individual metabolites and metabolic pathways associated with risk of developing PHN. The investigators hypothesize that alterations of plasma levels of certain metabolites and metabolic pathways previously implicated in chronic neuroimmune inflammation and increased neurosensitivity, including abnormal fatty acid and amino acid metabolism (e.g. arachidonic acid derived eicosanoids, glutamate-aspartate, tryptophan-kynurenine, and arginine-ornithine metabolic pathways), are involved in the development of PHN among women with HZ.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the NHS I, NHS II or HPFS cohort studies (n ~290,000)
* Provided information on weight and height at least one time
* Responded to at least one biennial questionnaire that included questions about HZ
* For the analyses examining obesity and risk of PHN, only participants in NHS I and NHS II who completed the ZSQ will be included

Exclusion Criteria:

* Reported date of HZ occurred before the study baseline
* Date of HZ cannot be determined
* Exposure information not available for the specific analysis

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Objective 1a: All participants from the NHS I, NHS II and HPFS (n ~209,000) who were enrolled at baseline and responded to a questionnaire that asked about HZ will be considered for inclusion.
  Objective 1b: All participants from the NHS I, NHS II and HPFS for whom plasma biomarker information is available will be considered for inclusion (n > 19,000).
  Objective 1c: All NHS I and NHS II participants who completed the Zoster Supplemental Questionnaire (ZSQ) and for whom information on metabolomics information is available will be considered for inclusion (n=1,005 to date).
  Objective 2a: All participants from the NHS I, NHS II and HPFS for whom we have comprehensive information on plasma metabolomics profiles (n >13,000) will be considered for inclusion.
  Objective 2b: All NHS I and NHS II participants who completed the ZSQ and for whom information on metabolomics information is available will be considered for inclusion (n=1,005 to date).
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 1976-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incident herpes zoster assessed by questionnaire | 2000-2024
  Biennial Questionnaires We have collected information about HZ and date of diagnosis on validated biennial questionnaires in the NHS I, NHS II and HPFS. These questionnaires were completed by over 200,000 participants. Participants were asked about clinician-diagnosed "shingles" and the year of diagnosis. We used the term "shingles" as this is the more commonly used name for HZ and to avoid confusion with other herpes virus infections. Over 30,000 cases of HZ have been reported. The validity of the self-reported HZ information was demonstrated by comparing reports of HZ by questionnaire with medical records in the subset of participants for whom medical records were obtained. Only the first report of HZ will be included for each participant.

SECONDARY OUTCOMES:
Post-herpetic neuralgia assessed by questionnaire | 2000-2024
  We obtained detailed information on HZ course, complications, treatment and other related factors by creating and administering a Zoster Supplemental Questionnaire (ZSQ). We administered the ZSQ to those participants in the NHS I and NHS II who reported "shingles" on the main questionnaires. We did not administer the ZSQ in HPFS due to the advanced age and the limited number of currently surviving participants. Specific information collected on the development of PHN will be used to identify cases of PHN among participants with a history of HZ. The validity of the self-reported PH information was demonstrated by comparing self-reports of PHN with medical records from a randomly selected subsets of participants. Only the first report of PHN for each participant will be used.

IPD SHARING:
Plan to Share IPD: No
We have a process for sharing data using a data enclave. Interested individuals should contact us.